CLINICAL TRIAL: NCT05913297
Title: Quantitative Neuroradiological Assessment of the Airways, Cranial Base Foramina, and Posterior Cranial Fossae in Children with Chiari Malformation: Relationship with Sleep Disorders
Brief Title: Neuroradiology Assesses Chiari Malformation's Impact on Airways, Cranial Base, and Sleep Disorders in Children.
Acronym: CHDSB
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Calandrelli Rosalinda, Principal Investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 5791 NO PROFIT
Record Dates: First submitted 2023-06-08; First posted 2023-06-22 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2024-06

CONDITIONS: Malformation Brain
MeSH Terms: interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Malformation Chiari 1: Magnetic Resonance
  Interventions: Diagnostic Test: Magnetic Resonance; Diagnostic Test: Polysomnographic evaluation
- Malformation Chiari 2: Magnetic Resonance
  Interventions: Diagnostic Test: Magnetic Resonance; Diagnostic Test: Polysomnographic evaluation

INTERVENTIONS:
Diagnostic Test: Magnetic Resonance — Magnetic Resonance
Diagnostic Test: Polysomnographic evaluation — Polysomnographic evaluation

SUMMARY:
The severity of sleep disorders in patients with Chiari malformations can vary. The investigators propose to establish a correlation between the severity of sleep-disordered breathing (SDB) and the quantitative neuroradiological data of the airways, cranial base foramina, and posterior cranial fossae

DETAILED DESCRIPTION:
Primary objective of the study is the evaluation of sleep-disordered breathing (SDB) in two distinct pediatric populations of patients with Chiari Malformation Type 1 (CM-I) and Chiari Malformation Type 2 (CM-II).

Secondary objectives:

Stratify the presence of SDB into central and obstructive origins in the two study populations.

Assess the volume of posterior cranial fossae, airway volume, and area of cranial base foramina in both groups.

Determine the relationships between SDB and morphological-quantitative anomalies associated with CM.

ELIGIBILITY:
Inclusion Criteria:

* Children (males or females) aged between 3 years and 18 years.
* Clinical diagnosis of Chiari malformation 1 and 2.
* Presence of informed consent for the initial clinical evaluation. The investigators commit to providing appropriate informational sheets to the parents of the patients (for those included in the study) during the initial clinical evaluation.

Exclusion Criteria:

* Chiari Malformation I and II associated with neurological diseases or craniofacial malformations.
* Cranial trauma or cardiac arrest.
* Administration of centrally acting medications within 2 weeks prior to the study, except for antiepileptic treatment for patients who have had seizures.
* Associated brain and cranial base tumors.
* Refusal to sign the informed consent for the initial clinical evaluation. The investigators commit to providing appropriate informational sheets to the parents of the patients (for those included in the study) during the initial clinical evaluation.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children (males or females) aged between 3 years and 18 years. Clinical diagnosis of Chiari malformation 1 and 2.
Sampling Method: Non-Probability Sample
Enrollment: 138 (Estimated)
Dates: Start 2023-06-08 (Actual); Primary Completion 2025-06-08 (Estimated); Study Completion 2026-06-08 (Estimated)

PRIMARY OUTCOMES:
prevalence of SDB | 3 years
  The primary endpoint of the study is the prevalence of sleep-disordered breathing (SDB) in two distinct pediatric populations of patients with CM-I and CM-II.

SECONDARY OUTCOMES:
volume of posterior cranial fossae | 3 years
  Evaluation of the volume of posterior cranial fossae CM-1 and CM-2, respectively, compared to an age-matched control group.
airway volume | 3 years
  Evaluation of the airway volume, in CM-1 and CM-2, respectively, compared to an age-matched control group
area of cranial base foramina | 3 years
  Evaluation of the area of cranial base foramina in CM-1 and CM-2, respectively, compared to an age-matched control group

CONTACTS AND LOCATIONS:
Overall Officials: Rosalinda Calandrelli, MD, Principal Investigator — Fondazione Policlinico A. Gemelli IRCCS
Locations (1):
- Fondazione Policlinico Gemelli IRCCS, Rome, Italy, Italy

IPD SHARING:
Plan to Share IPD: No